CLINICAL TRIAL: NCT05143541
Title: Use of a New Stapling Device in General Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Lexington Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Endostapler04
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2021-11

CONDITIONS: Thoracic Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- AEON Endostapler: Stapling performed with AEON Endostapler
  Interventions: Device: AEON Endostapler

INTERVENTIONS:
Device: AEON Endostapler — Surgery with AEON Endostapler

SUMMARY:
The goal of this study was to test the safety and efficacy of this stapler in our general thoracic surgery practice.

DETAILED DESCRIPTION:
A prospective study was conducted with 80 consecutive thoracic cases. Stapler usage data, intraoperative outcomes, and 30-day post-operative outcomes were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned VATS or open lung resection surgery (lobectomy or wedge resection)

Exclusion Criteria:

* Active bacterial or fungal infection
* Prior history of VATS or open lung surgery
* Use of staple line reinforcement material (buttress)
* Patients under the age of 18 on the date of the surgery
* Any female patient who is pregnant
* Scheduled concurrent surgical procedure other than lobectomy or wedge resection (central venous access - e.g., port placement, mediastinoscopy with lymph node sampling, and VATS lymphadenectomy are allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 subjects meeting inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AEON Endostapler
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Product Malfunction
Description: Number of participants with product malfunction. Product malfunction means any occurrence during the surgery where the stapler does not perform as intended.
Time Frame: Within surgery, up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
Participants | 0

2. Primary Outcome: Number of Participants With Intraoperative Staple Line Bleeding
Description: Number of participants with intraoperative staple line bleeding
Time Frame: Within surgery, up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
Participants | 0

3. Primary Outcome: Number of Participants With Reported Device-related Adverse Events
Description: Number of participants with reported device-related adverse events
Time Frame: Within 30-day post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
Participants | 0

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay (days)
Time Frame: Following hospital admission, up to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
days | 3.8 (3.2)

5. Secondary Outcome: Chest Tube Removal
Description: Time before chest tube removal (days)
Time Frame: Following surgery, up to chest tube removal
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AEON Endostapler
Number analyzed (Participants) | 80
days | 2.1 (2.7)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | AEON Endostapler
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT05143541/Prot_SAP_001.pdf